CLINICAL TRIAL: NCT00865787
Title: Effects of EGCG-Enhanced Extra Virgin Olive Oil on Endothelial Function
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Olivi Agri Team Srl- Grosetto, Italy (Unknown); University of Florence (Other)
Responsible Party: Amir Lerman, MN, Mayo Clinic
Other Study IDs: 07-002656
Record Dates: First submitted 2008-02-29; First posted 2009-03-19 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Olive Oil A
- Olive Oil B

SUMMARY:
This study is being done to determine if the use of EGCG-Enhanced Extra Virgin Olive Oil in a daily diet will improve endothelial function.

DETAILED DESCRIPTION:
Patients will be randomized to receive either placebo ROO (refined olive oil) or study solution EGCG-EVOO (EGCG enhanced extra-virgin olive oil) over the four month study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study if they have an abnormal endothelial function study. This is defined at our institution as an RH-PAT index of less than 2. Patients will undergo two RH-PAT analyses and included abnormal values are obtained on either one or both tests. Only patients who provide written informed consent will be included.

Exclusion Criteria:

* Patients with normal baseline endothelial function studies defined as RH-PAT index >2 will be excluded. Patients with uncontrolled hypertension >180/100 while on medication on initial evaluation will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic Patients
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Supplementation with enhanced olive oil will improve endothelial function as assessed by the reactive hyperemia peripheral arterial tonometry (RH-PAT) in patients with coronary artery disease (CAD) risk factors and endothelial dysfunction | Baseline and post 4 month

SECONDARY OUTCOMES:
Supplementation of EGCG enhanced olive oil will reduce peripheral markers of endothelial dysfunction and inflammation, oxidative stress and inflammation | Baseline and post 4 month

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- St Marys Hospital, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Widmer RJ, Freund MA, Flammer AJ, Sexton J, Lennon R, Romani A, Mulinacci N, Vinceri FF, Lerman LO, Lerman A. Beneficial effects of polyphenol-rich olive oil in patients with early atherosclerosis. Eur J Nutr. 2013 Apr;52(3):1223-31. doi: 10.1007/s00394-012-0433-2. Epub 2012 Aug 8. PMID 22872323